CLINICAL TRIAL: NCT03526991
Title: Exploring the Effects of Spinal Cord Stimulation in Parkinson's Disease.
Acronym: SCS for FOG
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Nora Vanegas (Other)
Responsible Party: Sponsor-Investigator, Nora Vanegas, Associate Professor of Neurology, Baylor College of Medicine
Organization: Baylor College of Medicine (Other)
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Device Feasibility
Other Study IDs: H-49023
Record Dates: First submitted 2018-05-04; First posted 2018-05-16 (Actual); Last update posted 2024-03-15 (Actual); Status verified 2024-03

CONDITIONS: Parkinson Disease
Keywords: Freezing of Gait; Locomotion; Spinal cord stimulation
MeSH Terms: conditions — Parkinson Disease

STUDY DESIGN:
Intervention Model Description: A total of 10 patients with a diagnosis of Parkinson's disease and treatment refractory freezing of gait will be recruited in this study.
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (2):
- Spinal Cord Stimulation (SCS) Tonic stimulation (Experimental): Tonic stimulation
  Interventions: Device: Spinal Cord Stimulator (SCS)
- Spinal Cord Stimulation (SCS) Burst stimulation (Experimental): Burst stimulation.
  Interventions: Device: Spinal Cord Stimulator (SCS)

INTERVENTIONS:
Device: Spinal Cord Stimulator (SCS) — The SCS implantation technique consists of inserting epidural leads-containing multiple stimulating electrodes (8). Two leads will be implanted percutaneously into the epidural space.
  The implantable pulse generator (IPG) is a neurostimulation system designed to deliver low-intensity electrical impulses. The system is intended to be used with leads and extensions that are compatible with the system. This neurostimulation system is indicated (FDA approved) as an aid in the management of chronic, intractable pain of the trunk and/or limbs. The intended use in this study is considered experimental.
  Other Names: Proclaim™ Implantable Pulse Generator with leads

SUMMARY:
Parkinson Disease (PD) patients experience a variety of motor issues such as walking difficulties, loss of balance, and freezing while walking, which impacts their quality of life. Some symptoms, like freezing of gait (FOG), do not respond to medications typically used to treat PD. Current surgical procedures used to alleviate PD symptoms also do not always improve FOG. Since many traditional therapies have failed for the treatment of FOG, researchers have proposed the use of newer treatments. Recent research in animal models and clinical human data using SCS has produced promising results, specifically showing improvement in FOG with the use of SCS in patients with PD.

The purpose of this study is to evaluate the effectiveness of spinal cord stimulation (SCS) for the management of freezing of gait (FOG) that does not respond to conventional treatments in subjects with Parkinson's disease (PD). The investigators hypothesize that SCS significantly decreases FOG episodes in patients with PD.

1. Assess the safety, tolerability and preliminary evidence of effectiveness of upper thoracic spinal cord stimulation for freezing of gait in Parkinson's (PD) patients.
2. Explore the effects of two SCS programming paradigms on motor, nonmotor and quality of life measures in PD patients with freezing of gait.

DETAILED DESCRIPTION:
Freezing of gait (FOG) is a devastating motor phenomenon which may occur in patients with Parkinson's Disease (PD) and other neurodegenerative disorders. It is characterized by episodes during which patients cannot generate effective forward stepping movements in the absence of motor deficits.

FOG leads to reduced mobility, loss of independence, social embarrassment, and caregiver stress. While most motor features of PD respond robustly to dopaminergic agents and deep brain stimulation (DBS), there are currently no effective treatments for FOG.

Indirect evidence from case reports of PD patients undergoing spinal cord stimulation (SCS) for neuropathic pain, has consistently described a positive effect of SCS on FOG. In addition, two recent reports demonstrated that thoracic SCS improved locomotion and FOG in patients with advanced PD. The promising role of SCS for the treatment of FOG in PD has encouraged us to assemble a multi-disciplinary team for the systematic investigation of the motor effects of SCS on FOG, locomotion and other parkinsonian features.

The current study integrates minimally invasive SCS and the use of robotic technology to determine objective gait parameters. The investigators propose a pilot study for the implantation of SCS to the spinal cord on PD patients with treatment-refractory FOG, including a longitudinal assessment of motor outcomes. Motors assessments will include: PAMSys and LEGSys to characterize gait, ActivePERS motion sensor to monitor ambulation parameters and overall activity at home, participants will also be given electronic tablets for the ActivePERS to collect real time information about falls.

ELIGIBILITY:
Inclusion Criteria:

* Males and females between older than 18 years of age.
* Able to provide informed consent
* Diagnosed with idiopathic PD (meeting at least two of the three United Kingdom (UK) Brain Bank criteria for PD, specifically bradykinesia plus resting tremor or rigidity) whose major complaints is levodopa refractory FOG. Levodopa refractoriness will be defined as lack of subjective improvement on FOG episodes as reported by the patient.
* Documented dopaminergic response
* Optimized PD treatment including dopaminergic medications, and/or deep brain stimulation (DBS) therapy
* Presence of at least two self-reported levodopa refractory episodes of FOG per day, not limited to start hesitation
* At least one witnessed freezing event during the screening visit in the 'on' medication state (defined as 45 minutes after a regular dose of Levodopa for the subject being studied)

Exclusion Criteria:

Presence of any co-morbid psychiatric illness(es) that would interfere with the completion of the study or pose risk to the patient, as defined below:

* Presence of psychosis
* Depression BDI >14
* Anxiety BAI >14

  * Presence of an active infection, uncontrolled diabetes mellitus, immunosuppression or other medical contraindications to undergoing SCS implantation
  * Patients who are currently on anticoagulation treatment or unable to hold off the anticoagulants (including Plavix, Aspirin, Warfarin, etc.) 7 days prior to the SCS procedure.
  * Moderate Cognitive Impairment defined by a MoCA < 23
  * Diagnosis of failed back surgery syndrome, Complex Regional Pain Syndrome (CRPS) or intractable low back pain and leg pain.
  * Women of childbearing potential will be excluded as from participation due to the limited safety data of thoracic SCS on the fetus.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Estimated)
Dates: Start 2021-08-01 (Actual); Primary Completion 2025-06-30 (Estimated); Study Completion 2025-06-30 (Estimated)

PRIMARY OUTCOMES:
Safety and Tolerability | 12-months
  Incidence of Adverse Events as assessed by Adverse Event reporting.

SECONDARY OUTCOMES:
Change in New Freezing of Gait Questionnaire (NFOG-Q) score | Baseline (pre-surgery), and over a 12month follow up period
  The New Freezing of Gait Questionnaire (NFOG-Q) is a clinician-administered tool that aims to assess both the clinical aspects of FOG as well as its subsequent impairments on quality of life. The task ratings and scales are calculated into a summed NFOG-Q score. The scale is scored from 0-28. A score of 0 means least severe. A score of 28 means the most severe.
10-meter walk | Baseline (pre-surgery), and over a 12-month follow up period
  The 10-meter walk measures gait velocity. The 10-meter walk is measured in the length of time duration taken to complete. A lower duration means a higher gait speed. A high duration means a lower gain speed.
Montreal Cognitive Assessment (MoCA), | Baseline (pre-surgery), and over a 12month follow up period
  This is a test of cognitive function used to screen and track cognitive changes over time. The MoCA is scored between 0 - 30 which 0 meaning there is an abnormal amount of cognitive function and 30 meaning there is a normal amount of cognitive function.
Change in MDS-UPDRS score | Baseline (pre-surgery), and over a 12month follow up period
  The Movement Disorder Society (MDS) published a revision of the unified Parkinson's disease rating scale, known as the MDS-UPDRS. The Part III: Motor Examination portion of the scale assesses the motor signs of PD and is completed by the examiner. The measure is scored between 0 - 76 with 0 have the most abnormal motor signs and 76 having normal motor signs.
Non-Motor Symptoms Scale (NMSS) | Baseline (pre-surgery), and over a 12month follow up period
  Symptoms assessed over the last month. Each symptom scored with respect to: Severity: 0 = None, 1 = Mild: symptoms present but causes little distress or disturbance to patient; 2 = Moderate: some distress or disturbance to patient; 3 = Severe: major source of distress or disturbance to patient. The measure is scored between 0 - 360, with 0 meaning there are no non-motor symptoms and 360 meaning there are non-motor symptoms.
Parkinson's Disease Questionnaire (PDQ39) | Baseline (pre-surgery), and over a 12month follow up period
  The PDQ-39 is a 39-item self-report questionnaire, which assesses Parkinson's disease-specific health related quality of life. The measure is scored between 0 - 100 with 0 meaning no health problems and 100 meaning more health problems.

CONTACTS AND LOCATIONS:
Overall Officials: Nora Vanegas, MD, Principal Investigator — Baylor College of Medicine
Locations (2):
- United States (2):
  - Columbia University, New York, New York
  - Baylor College of Medicine, Houston, Texas

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Giladi N, Kao R, Fahn S. Freezing phenomenon in patients with parkinsonian syndromes. Mov Disord. 1997 May;12(3):302-5. doi: 10.1002/mds.870120307. PMID 9159723
- [Background] Schoneburg B, Mancini M, Horak F, Nutt JG. Framework for understanding balance dysfunction in Parkinson's disease. Mov Disord. 2013 Sep 15;28(11):1474-82. doi: 10.1002/mds.25613. Epub 2013 Aug 7. PMID 23925954
- [Background] Espay AJ, Fasano A, van Nuenen BF, Payne MM, Snijders AH, Bloem BR. "On" state freezing of gait in Parkinson disease: a paradoxical levodopa-induced complication. Neurology. 2012 Feb 14;78(7):454-7. doi: 10.1212/WNL.0b013e3182477ec0. Epub 2012 Jan 18. PMID 22262741
- [Background] Fasano A, Lozano AM. Deep brain stimulation for movement disorders: 2015 and beyond. Curr Opin Neurol. 2015 Aug;28(4):423-36. doi: 10.1097/WCO.0000000000000226. PMID 26110808
- [Background] Fenelon G, Goujon C, Gurruchaga JM, Cesaro P, Jarraya B, Palfi S, Lefaucheur JP. Spinal cord stimulation for chronic pain improved motor function in a patient with Parkinson's disease. Parkinsonism Relat Disord. 2012 Feb;18(2):213-4. doi: 10.1016/j.parkreldis.2011.07.015. Epub 2011 Aug 23. No abstract available. PMID 21865071
- [Background] Soltani F, Lalkhen A. Improvement of Parkinsonian Symptoms With Spinal Cord Stimulation: Consequence or Coincidence? J Neurol Neurosurg Psychiatry. 2013;84(11):e2.74-e2. doi:10.1136/jnnp-2013-306573.165.
- [Background] Hassan S, Amer S, Alwaki A, Elborno A. A patient with Parkinson's disease benefits from spinal cord stimulation. J Clin Neurosci. 2013 Aug;20(8):1155-6. doi: 10.1016/j.jocn.2012.08.018. Epub 2013 Feb 26. PMID 23453160
- [Background] Pinto de Souza C, Hamani C, Oliveira Souza C, Lopez Contreras WO, Dos Santos Ghilardi MG, Cury RG, Reis Barbosa E, Jacobsen Teixeira M, Talamoni Fonoff E. Spinal cord stimulation improves gait in patients with Parkinson's disease previously treated with deep brain stimulation. Mov Disord. 2017 Feb;32(2):278-282. doi: 10.1002/mds.26850. Epub 2016 Nov 10. PMID 27862267
- [Background] Rohani M, Kalsi-Ryan S, Lozano AM, Fasano A. Spinal cord stimulation in primary progressive freezing of gait. Mov Disord. 2017 Sep;32(9):1336-1337. doi: 10.1002/mds.27103. Epub 2017 Jul 6. No abstract available. PMID 28681922
- [Background] Giladi N, Tal J, Azulay T, Rascol O, Brooks DJ, Melamed E, Oertel W, Poewe WH, Stocchi F, Tolosa E. Validation of the freezing of gait questionnaire in patients with Parkinson's disease. Mov Disord. 2009 Apr 15;24(5):655-61. doi: 10.1002/mds.21745. PMID 19127595
- [Background] de Lau LM, Breteler MM. Epidemiology of Parkinson's disease. Lancet Neurol. 2006 Jun;5(6):525-35. doi: 10.1016/S1474-4422(06)70471-9. PMID 16713924
- [Background] Shulman JM, De Jager PL, Feany MB. Parkinson's disease: genetics and pathogenesis. Annu Rev Pathol. 2011;6:193-222. doi: 10.1146/annurev-pathol-011110-130242. PMID 21034221
- [Background] Turner BM, Forstmann BU, Love BC, Palmeri TJ, Van Maanen L. Approaches to Analysis in Model-based Cognitive Neuroscience. J Math Psychol. 2017 Feb;76(B):65-79. doi: 10.1016/j.jmp.2016.01.001. Epub 2016 Feb 17. PMID 31745373
- [Background] Snijders AH, Takakusaki K, Debu B, Lozano AM, Krishna V, Fasano A, Aziz TZ, Papa SM, Factor SA, Hallett M. Physiology of freezing of gait. Ann Neurol. 2016 Nov;80(5):644-659. doi: 10.1002/ana.24778. Epub 2016 Oct 7. PMID 27649270
- [Background] Fleury V, Pollak P, Gere J, Tommasi G, Romito L, Combescure C, Bardinet E, Chabardes S, Momjian S, Krainik A, Burkhard P, Yelnik J, Krack P. Subthalamic stimulation may inhibit the beneficial effects of levodopa on akinesia and gait. Mov Disord. 2016 Sep;31(9):1389-97. doi: 10.1002/mds.26545. Epub 2016 Feb 17. PMID 26887333
- [Background] Adams C, Keep M, Martin K, McVicker J, Kumar R. Acute induction of levodopa-resistant freezing of gait upon subthalamic nucleus electrode implantation. Parkinsonism Relat Disord. 2011 Jul;17(6):488-90. doi: 10.1016/j.parkreldis.2011.02.014. Epub 2011 Mar 11. No abstract available. PMID 21397548
- [Background] van Nuenen BF, Esselink RA, Munneke M, Speelman JD, van Laar T, Bloem BR. Postoperative gait deterioration after bilateral subthalamic nucleus stimulation in Parkinson's disease. Mov Disord. 2008 Dec 15;23(16):2404-6. doi: 10.1002/mds.21986. PMID 18951532
- [Background] Rocchi L, Carlson-Kuhta P, Chiari L, Burchiel KJ, Hogarth P, Horak FB. Effects of deep brain stimulation in the subthalamic nucleus or globus pallidus internus on step initiation in Parkinson disease: laboratory investigation. J Neurosurg. 2012 Dec;117(6):1141-9. doi: 10.3171/2012.8.JNS112006. Epub 2012 Oct 5. PMID 23039143
- [Background] Ferraye MU, Debu B, Fraix V, Goetz L, Ardouin C, Yelnik J, Henry-Lagrange C, Seigneuret E, Piallat B, Krack P, Le Bas JF, Benabid AL, Chabardes S, Pollak P. Effects of pedunculopontine nucleus area stimulation on gait disorders in Parkinson's disease. Brain. 2010 Jan;133(Pt 1):205-14. doi: 10.1093/brain/awp229. Epub 2009 Sep 22. PMID 19773356
- [Background] Thevathasan W, Cole MH, Graepel CL, Hyam JA, Jenkinson N, Brittain JS, Coyne TJ, Silburn PA, Aziz TZ, Kerr G, Brown P. A spatiotemporal analysis of gait freezing and the impact of pedunculopontine nucleus stimulation. Brain. 2012 May;135(Pt 5):1446-54. doi: 10.1093/brain/aws039. Epub 2012 Mar 6. PMID 22396391
- [Background] Zrinzo L, Zrinzo LV, Hariz M. The peripeduncular nucleus: a novel target for deep brain stimulation? Neuroreport. 2007 Aug 6;18(12):1301-2. doi: 10.1097/WNR.0b013e3282638603. PMID 17632287
- [Background] Thevathasan W, Coyne TJ, Hyam JA, Kerr G, Jenkinson N, Aziz TZ, Silburn PA. Pedunculopontine nucleus stimulation improves gait freezing in Parkinson disease. Neurosurgery. 2011 Dec;69(6):1248-53; discussion 1254. doi: 10.1227/NEU.0b013e31822b6f71. PMID 21725254
- [Background] Compton AK, Shah B, Hayek SM. Spinal cord stimulation: a review. Curr Pain Headache Rep. 2012 Feb;16(1):35-42. doi: 10.1007/s11916-011-0238-7. PMID 22086473
- [Background] Fuentes R, Petersson P, Siesser WB, Caron MG, Nicolelis MA. Spinal cord stimulation restores locomotion in animal models of Parkinson's disease. Science. 2009 Mar 20;323(5921):1578-82. doi: 10.1126/science.1164901. PMID 19299613
- [Background] Shealy CN, Mortimer JT, Reswick JB. Electrical inhibition of pain by stimulation of the dorsal columns: preliminary clinical report. Anesth Analg. 1967 Jul-Aug;46(4):489-91. No abstract available. PMID 4952225
- [Background] Cook AW, Weinstein SP. Chronic dorsal column stimulation in multiple sclerosis. Preliminary report. N Y State J Med. 1973 Dec 15;73(24):2868-72. No abstract available. PMID 4543587
- [Background] Thiriez C, Gurruchaga JM, Goujon C, Fenelon G, Palfi S. Spinal stimulation for movement disorders. Neurotherapeutics. 2014 Jul;11(3):543-52. doi: 10.1007/s13311-014-0291-0. PMID 25015323
- [Background] Thevathasan W, Mazzone P, Jha A, Djamshidian A, Dileone M, Di Lazzaro V, Brown P. Spinal cord stimulation failed to relieve akinesia or restore locomotion in Parkinson disease. Neurology. 2010 Apr 20;74(16):1325-7. doi: 10.1212/WNL.0b013e3181d9ed58. No abstract available. PMID 20404313
- [Background] Santana MB, Halje P, Simplicio H, Richter U, Freire MAM, Petersson P, Fuentes R, Nicolelis MAL. Spinal cord stimulation alleviates motor deficits in a primate model of Parkinson disease. Neuron. 2014 Nov 19;84(4):716-722. doi: 10.1016/j.neuron.2014.08.061. Epub 2014 Oct 30. PMID 25447740
- [Background] Agari T, Date I. Spinal cord stimulation for the treatment of abnormal posture and gait disorder in patients with Parkinson's disease. Neurol Med Chir (Tokyo). 2012;52(7):470-4. doi: 10.2176/nmc.52.470. PMID 22850494
- [Background] Kiriakopoulos ET, Tasker RR, Nicosia S, Wood ML, Mikulis DJ. Functional magnetic resonance imaging: a potential tool for the evaluation of spinal cord stimulation: technical case report. Neurosurgery. 1997 Aug;41(2):501-4. doi: 10.1097/00006123-199708000-00042. PMID 9257323
- [Background] Holsheimer J. Which Neuronal Elements are Activated Directly by Spinal Cord Stimulation. Neuromodulation. 2002 Jan;5(1):25-31. doi: 10.1046/j.1525-1403.2002._2005.x. PMID 22151778
- [Background] Weise D, Winkler D, Meixensberger J, Classen J. Effects of spinal cord stimulation in a patient with Parkinson's disease and chronic back pain. J Neurol. 2010;257:S217.
- [Background] Yadav AP, Nicolelis MAL. Electrical stimulation of the dorsal columns of the spinal cord for Parkinson's disease. Mov Disord. 2017 Jun;32(6):820-832. doi: 10.1002/mds.27033. Epub 2017 May 12. PMID 28497877
- [Background] Gazelka HM, Freeman ED, Hooten WM, Eldrige JS, Hoelzer BC, Mauck WD, Moeschler SM, Pingree MJ, Rho RH, Lamer TJ. Incidence of clinically significant percutaneous spinal cord stimulator lead migration. Neuromodulation. 2015 Feb;18(2):123-5; discussion 125. doi: 10.1111/ner.12184. Epub 2014 May 5. PMID 24796230
- [Background] Hoelzer BC, Bendel MA, Deer TR, Eldrige JS, Walega DR, Wang Z, Costandi S, Azer G, Qu W, Falowski SM, Neuman SA, Moeschler SM, Wassef C, Kim C, Niazi T, Saifullah T, Yee B, Kim C, Oryhan CL, Rosenow JM, Warren DT, Lerman I, Mora R, Hayek SM, Hanes M, Simopoulos T, Sharma S, Gilligan C, Grace W, Ade T, Mekhail NA, Hunter JP, Choi D, Choi DY. Spinal Cord Stimulator Implant Infection Rates and Risk Factors: A Multicenter Retrospective Study. Neuromodulation. 2017 Aug;20(6):558-562. doi: 10.1111/ner.12609. Epub 2017 May 11. PMID 28493599
- [Background] Mekhail NA, Mathews M, Nageeb F, Guirguis M, Mekhail MN, Cheng J. Retrospective review of 707 cases of spinal cord stimulation: indications and complications. Pain Pract. 2011 Mar-Apr;11(2):148-53. doi: 10.1111/j.1533-2500.2010.00407.x. Epub 2010 Sep 8. PMID 21371254
- [Background] Engle MP, Vinh BP, Harun N, Koyyalagunta D. Infectious complications related to intrathecal drug delivery system and spinal cord stimulator system implantations at a comprehensive cancer pain center. Pain Physician. 2013 May-Jun;16(3):251-7. PMID 23703411
- [Background] Turner JA, Loeser JD, Deyo RA, Sanders SB. Spinal cord stimulation for patients with failed back surgery syndrome or complex regional pain syndrome: a systematic review of effectiveness and complications. Pain. 2004 Mar;108(1-2):137-47. doi: 10.1016/j.pain.2003.12.016. PMID 15109517
- [Background] Minto S, Zanotto D, Boggs EM, Rosati G, Agrawal SK. Validation of a Footwear-Based Gait Analysis System With Action-Related Feedback. IEEE Trans Neural Syst Rehabil Eng. 2016 Sep;24(9):971-980. doi: 10.1109/TNSRE.2015.2498287. Epub 2015 Nov 5. PMID 26561476
- [Background] Nieuwboer A, Rochester L, Herman T, Vandenberghe W, Emil GE, Thomaes T, Giladi N. Reliability of the new freezing of gait questionnaire: agreement between patients with Parkinson's disease and their carers. Gait Posture. 2009 Nov;30(4):459-63. doi: 10.1016/j.gaitpost.2009.07.108. Epub 2009 Aug 5. PMID 19660949